CLINICAL TRIAL: NCT00649246
Title: 1. Prospective Studies in Infants of the Immunopathogenesis of Type 1 Diabetes 2. Consortium for Identification of Environmental Triggers of Type 1 Diabetes: MCG/UF Clinical Center 3. Identification of Serum Protein Markers for Type 1 Diabetes Using Mass-Spectrometry Techniques 4. Validation of Microarray-Based Biomarkers for Type 1 Diabetes 5. Development of Microarray-Based Biomarkers for Type 1 Diabetes 6. Proteomic Changes/Progression of Human Type 1 Diabetes 7. Identification and Validation of Serum Biomarkers for T1D
Brief Title: Prospective Assessment in Newborns for Diabetes Autoimmunity
Acronym: PANDA
Status: Completed | Type: Observational
Sponsor: Augusta University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); University of Florida (Other); Emory University (Other); Medical University of South Carolina (Other); University of South Carolina (Other)
Responsible Party: Principal Investigator, Jin-Xiong She, Director Center for Biotechnology and Genomic Medicine, Augusta University
Other Study IDs: DK63865 - PANDA; U01DK063865 (NIH)
Record Dates: First submitted 2008-03-28; First posted 2008-04-01 (Estimated); Last update posted 2018-03-27 (Actual); Status verified 2018-03

CONDITIONS: Type 1 Diabetes; Autoimmunity
Keywords: genetics; type 1 diabetes; biomarkers; autoimmunity
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Autoimmune Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood, DNA, serum, RNA, urine
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- 1: controls:
  healthy individuals with no family history of type 1 diabetes
- 2: high-risk:
  Subjects with islet autoantibodies or high-risk diabetes genes
- 3: type 1 diabetes:
  subjects with type 1 diabetes

SUMMARY:
This is an observational study designed to help researchers understand the genetics and pathogenesis of type 1 diabetes, and to identify biomarkers for disease and disease complication prediction.

DETAILED DESCRIPTION:
This study is designed to identify people who are at risk for developing type 1 diabetes, based on their genetics, family history and autoimmunity status, and to understand the role genetics plays in the development of the complications associated with type 1 diabetes in patients already affected by type 1 diabetes.

ELIGIBILITY:
Inclusion Criteria: all are welcome -

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: newborns, young children, adults with or without type 1 diabetes
Sampling Method: Non-Probability Sample
Enrollment: 25055 (Actual)
Dates: Start 1997-07; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
autoantibodies against the pancreas and type 1 diabetes | 50 years

SECONDARY OUTCOMES:
Risk factors for type 1 diabetes | 50 years

CONTACTS AND LOCATIONS:
Overall Officials: Jin Xiong She, PhD, Principal Investigator — Augusta University
Locations (3):
- United States (3):
  - University of Florida, Gainesville, Florida
  - Medical University of South Carolina, Charleston, South Carolina
  - University of South Carolina, Columbia, South Carolina

REFERENCES:
- See also: PANDA web site — http://www.pandastudy.org